CLINICAL TRIAL: NCT01020344
Title: Randomized Controlled Trial on the Cardiovascular Effects of Lung Volume Reduction Surgery in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Mechanisms of Vascular Damage in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPD-CVD2
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung volume reduction surgery (Active Comparator): This group will receive lung volume reduction surgery
  Interventions: Procedure: Lung volume reduction surgery
- No lung volume reduction surgery (No Intervention): This group will not receive LVRS during the 3 months of the study

INTERVENTIONS:
Procedure: Lung volume reduction surgery — Lung volume reduction surgery
  Arms: Lung volume reduction surgery

SUMMARY:
A randomised controlled trial will be performed to evaluate the effects of lung volume reduction surgery (LVRS) in patients with COPD on systemic inflammation, oxidative stress, endothelial function, arterial stiffness and blood pressure. We hypothesize that LVRS will lead to a reduction of systemic inflammation, oxidative stress, arterial stiffness and blood pressure and to improved endothelial function.

For this purpose 30 patients with severe/very severe COPD (GOLD III-IV) and pulmonary emphysema who are to undergo LVRS will be randomised to one of two groups: group 1 receiving immediate LVRS and group 2 receiving LVRS after a delay of 3 months.

Measures of systemic inflammation, oxidative stress, endothelial function, arterial stiffness and blood pressure will be measured at baseline and 3 months after surgery and no surgery, respectively (group 2 receiving surgery only after a delay of 3 months will serve as control group) to investigate the effects of LVRS on the described outcomes.

DETAILED DESCRIPTION:
Not desired

ELIGIBILITY:
Inclusion criteria:

* Dyspnea at rest or at minimal physical activity, severe limitation of exercise capacity (6-min walk distance < 350 m).
* Acceptance of an increased perioperative mortality (approximately 2 %) and/or morbidity (long lasting hospitalization due to prolonged air leaks)
* COPD (GOLD guidelines) with severe obstructive ventilatory defect (FEV1 <35% predicted)
* Functional aspects of lung emphysema, i.e. irreversible hyperinflation with a residual volume to total lung capacity ratio (RV/TLC) of >0.65 and an impaired total lung diffusion capacity (DLCO), usually < 40% predicted.
* Pulmonary emphysema confirmed by high resolution computer tomography

Exclusion criteria: - Current smokers

* Age > 75years
* "Vanishing" lung or diffuse lung emphysema on CT, FEV1 <20% predicted and DLCO <20% predicted, and hypercapnia (PaCO2 >7.3kPa)
* Overt active coronary artery disease, severe left ventricular function impairment
* Pulmonary hypertension with a mean pulmonary artery pressure >35 mmHg at rest
* Acute bronchopulmonary infection, bronchiectasis on high resolution tomography
* Pulmonary cachexia (body mass index <18kg/m2)
* Neoplastic disease with a life expectancy of less than 2 years
* Addiction to alcohol/drugs
* Relevant renal (creatinine >150ug/ml), active gastroenterological (GI-bleeding in the previous year, abnormal liver function, active inflammatory bowel disease) or active neurological disease.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
1. Systemic inflammation 2. Vascular function | Before and 3 months after surgery/no surgery

SECONDARY OUTCOMES:
1. Oxidative stress 2. Blood pressure 3. Physical Activity 4. Lung function 5. Hypoxemia | Before and 3 months after surgery/no surgery

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Leading Physician, Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (1):
- Pulmonary Division, University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Clarenbach CF, Sievi NA, Brock M, Schneiter D, Weder W, Kohler M. Lung Volume Reduction Surgery and Improvement of Endothelial Function and Blood Pressure in Patients with Chronic Obstructive Pulmonary Disease. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2015 Aug 1;192(3):307-14. doi: 10.1164/rccm.201503-0453OC. PMID 26016823